CLINICAL TRIAL: NCT03470948
Title: Utility of Surgical Apgar Score in Predicting Post-Operative Complications After Whipple Procedure in Pancreatic Cancer Patients
Brief Title: Surgical Apgar Score After Whipple Procedure in Pancreatic Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: No manpower to conduct the study further
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Raghu Thota, Professor, Tata Memorial Hospital
Other Study IDs: TataMH
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Complications
Keywords: surgical apgar score, postoperative complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observe postoperative complications — The aim of this study is to confirm the utility of a 10-point Surgical Apgar Score to rate surgical outcomes in Whipples procedure in patients with pancreatic cancer.

SUMMARY:
The number of new cases of pancreatic cancer is 12.4 per 100,000 men and women per year. The number of deaths is 10.9 per 100,000 men and women per year. These rates are age-adjusted and based on 2009-2013 cases and deaths1. This cancer has a very poor prognosis and around 7.7% of these patients have a 5 years survival rate. Whipple procedure is the surgical treatment option for cancer pancreas, where the head of the pancreas, the gallbladder, part of the stomach, part of the small intestine, and the bile duct are removed.Those that undergoes this procedure, the 5 year survival rate increases to about 20%2. The duration of intensive care unit monitoring and hospital stay are longer than for most upper gastrointestinal surgeries. Pancreaticoduodenectomy is a major operation, carrying significant risk of morbidity and mortality with 30 - 60% complication rate3. The possibility of identifying patients at risk for postoperative complications and targeting them from surveillance and early treatment offers an opportunity to develop interventions that might significantly improve outcomes and efficiency. Gawande et al. developed and validated the surgical Apgar score (SAS) and demonstrated that SAS can be useful for rating the condition of patients after general or vascular surgery4. SAS is based on intraoperative blood loss, blood pressure, and heart rate3. The score is very simple and easy to calculate and can be available immediately after surgery. Several validation studies have reported that SAS is useful for predicting the risk of complications associated with various procedures4-10. We investigated this SAS could predict major postoperative complications among patients undergoing Whipples procedure in patients with pancreatic cancer.

DETAILED DESCRIPTION:
This is a prospective, observational, non-interventional, non-randomized study involving the adult patients undergoing Whipple's procedure. Institutional ethics permission and written informed consent will be taken from the patient. The study duration will be for a period of 5 years, but the data of the first one year will be analysed and will presented as a thesis for MD (Anaesthesia). Administration of anaesthesia and reversal of neuromuscular blocking drugs will be carried as per the institutional routine practice and at the discretion of anaesthesiologist in charge. The study will include patients undergoing Whipple's procedure for pancreatic cancer, between age group of 18-75years, with ASA-PS I - III. Preoperative, intraoperative and outcome variables as defined according to the definitions established by the American college of surgeons National Surgeons Quality Improvement Program (NSQIP) will be recorded. A total of 11 preoperative, 14 intraoperative and 21 outcome variables will be collected (see Appendix). All the post operative outcome variables will be defined. Preoperative comorbid conditions will also be recorded. SAS will be calculated from three intraoperative variables (1) the estimated blood loss (EBL), (2) lowest heart rate (HR), and (3) lowest mean arterial pressure (MAP). For analysis, SAS will be classified as low (≤ 4 points), intermediate (5-6 points) and high (7-9 points). Complications including mortality will be assessed Upto 30 days postoperatively. The categorization of the complications as major and minor is consistent with NSQIP definition. Major complications include acute kidney injury, blood loss ≥ 2000ml, transfusion requiring ≥ 4 U packed blood cells within 72 hours of surgery, cardiac or respiratory arrest requiring cardiopulmonary resuscitation (CPR), coma for 24 hours or longer, deep venous thrombosis, septic shock, acute myocardial infarction, new onset arrhythmias, unplanned re-intubation, ventilator use for 48 hours or longer, pneumonia, pulmonary embolism, stroke, wound disruption, deep or organ space surgical site infection, sepsis, systemic inflammatory response syndrome, unplanned intensive care unit (ICU) admission, need for reoperation, anastomotic leak or fistula, vascular, ureteral or neural injuries, unplanned readmission < 30 days of discharge, and death. The occurrence of major postoperative complications within 30 days of surgery represents primary outcome. Some of the patients do follow-up at day 30 to the OPD and those patients who don't follow-up at day 30 will be assessed and interviewed by telephone. If they are not able to follow-up on day 30, they will be contacted telephonically and interviewed for a period of 10-15 minutes, by a research nurse or a research doctor. Only mortality will be noted at day 30.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing Whipple's procedure for pancreatic cancer,
* between age group of 18-75years,
* with ASA-PS I - III.

Exclusion Criteria:

* Age <18 and >75yrs.
* Pt not consenting,
* ASA IV & above

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study to be done for a period of 60 months. Upto 750 patients in 60 months, thus 150 patients in 12 months
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of major postoperative complications and/or death within 30 days of surgery | 30 days postoperative
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Patil, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No